CLINICAL TRIAL: NCT03550898
Title: Can Dynamic Ultrasonography Replace Urodynamics in the Follow-up of Patients With Myelomeningocele: A Prospective Concurrent Study
Brief Title: Can Dynamic Ultrasonography Replace Urodynamics in Follow-up of Patients With Myelomeningocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 15-0287
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Neurogenic Bladder; Myelomeningocele
Keywords: Dynamic Ultrasonography; Spinal Dysraphism
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Meningomyelocele; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Dynamic ultrasonography was performed in all patients during the urodynamic study.
Masking Description: Dynamic ultrasonography was performed during the filling phase of the urodynamic study. The radiologist and the urodynamicist had no verbal or visual contact during the examinations, with use of a siding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic ultrasonography (Other): Dynamic ultrasonography was performed in all patients who underwent urodynamics, simultaneously.
  Interventions: Diagnostic Test: Dynamic Ultrasonography

INTERVENTIONS:
Diagnostic Test: Dynamic Ultrasonography — Dynamic Ultrasonography was performed with patients in supine position, with a suprapubic sagittal position transductor, during filling phase of urodynamics.

SUMMARY:
Patients with neurogenic bladder need periodic evaluation with urodynamic study, a invasive and uncomfortable procedure.

Aim: To evaluate the accuracy of dynamic ultrasonography as a feasible and noninvasive alternative diagnostic method to identify detrusor overactivity in patients with neurogenic bladder

DETAILED DESCRIPTION:
The urodynamic study and dynamic ultrasonography were performed concurrently, to identify detrusor overactivity, in patients with myelomeningocele and clinical indication for urodynamics, by investigators without verbal or visual contact.

The overactivity was diagnosed through active conformational change of the bladder during filling phase.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients of the Pediatric Urology Department of the investigator's institution with diagnosis of myelomeningocele and clinical indication for urodynamic study

Exclusion Criteria:

* Previous bladder augmentation surgery
* Current urinary tract infection
* Fail to provide consent for participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of dynamic ultrasonography to identify bladder overactivity in neurogenic bladder. | 20 minutes
  Dynamic Ultrasonography evaluated the dynamic conformational change of the bladder to identify the presence of detrusor overactivity, based on a subjective graduation of contractions, compared to the urodynamic data.

SECONDARY OUTCOMES:
To evaluate the accuracy of dynamic ultrasonography to identify maximum cystometric capacity. | 20 minutes
  The bladder maximum capacity was measured at the end of the filling phase, based on the ellipse formula and compared to the infused volume in urodynamics.
To assess the ability of dynamic ultrasonography to estimate the pressure of detrusor contractions. | 20 minutes
  According to the detrusor mobility and bladder deformity, the contractions were graded: 1 - no contractions; 2 - partial contraction of bladder floor; 3 - partial contraction of bladder floor and posterior wall; 4 - generalized contraction with modification of bladder shape from ellipsoid to round. These data were compared to the maximum pressure data recorded in the urodynamic study.

CONTACTS AND LOCATIONS:
Overall Officials: Brasil S Neto, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided